CLINICAL TRIAL: NCT02224560
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P; CBD) as Adjunctive Treatment for Seizures Associated With Lennox-Gastaut Syndrome in Children and Adults.
Brief Title: Efficacy and Safety of GWP42003-P for Seizures Associated With Lennox-Gastaut Syndrome in Children and Adults
Acronym: GWPCARE3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1414; 2014-002940-42 (EudraCT Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Lennox Gastaut Syndrome
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GWP42003-P 20 mg/kg/day Dose (Experimental): Participants received GWP42003-P 20 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P
- GWP42003-P 10 mg/kg/day Dose (Experimental): Participants received GWP42003-P 10 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 10 mg/kg/day over 7 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Participants received placebo (0 mg/mL CBD) volume matched to 1 of the 2 dose levels (10 or 20 mg/kg/day) administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 7 to 11 days according to the matched IMP group (7 or 11 days for the 10 or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period.
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: GWP42003-P — GWP42003-P was presented as an oral solution containing 100 mg/milliliter (mL) cannabidiol (CBD) in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL). Participants were randomly assigned to receive either 10 or 20 mg/kg/day.
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 10 mg/kg/day Dose; GWP42003-P 20 mg/kg/day Dose
Drug: Placebo control — Placebo was presented as an oral solution containing 0 mg/mL CBD in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the efficacy of GWP42003-P as adjunctive treatment in reducing the number of drop seizures when compared with placebo in participants with Lennox-Gastaut syndrome (LGS).

DETAILED DESCRIPTION:
This study was a 1:1:1 randomized, double-blind, 14-week comparison of 2 dose levels (10 milligram [mg] per kilogram [kg] per day [mg/kg/day] and 20 mg/kg/day) of GWP42003-P versus placebo. Participants who satisfied all inclusion and none of the exclusion criteria began a 28-day baseline observation period. The treatment period consisted of a 2-week titration period followed by a 12-week maintenance period. The 20 mg/kg/day dose was recommended by the Data Safety Monitoring Committee (DSMC) after assessment of safety and pharmacokinetic data from Part A of study GWEP1332 (NCT02091206). The 10 mg/kg/day dose was defined as 50% of the 20 mg/kg/day dose. The first participant was not enrolled into this study until the DSMC had reviewed the safety data from Part A of study GWEP1332.

Participants who satisfied all eligibility criteria were randomized at Day 1 to receive 10 mg/kg/day GWP42003-P, 20 mg/kg/day GWP42003-P, or placebo at a 1:1:1 ratio. Participants in the placebo group were split into 2 equivalent cohorts; one half received 10 mg/kg/day dosing volumes and one half received 20 mg/kg/day dosing volumes. The 2 placebo cohorts were pooled for the analyses of efficacy. Participants titrated GWP42003-P to the 10 mg/kg/day or 20 mg/kg/day (or equivalent volume of placebo) dose over 7 and 11 days, respectively, and remained at this dose for the 12-week maintenance period. Following the end of treatment (Day 99), participants were invited to continue to receive GWP42003-P in an open-label extension (OLE) study under a separate protocol (GWEP1415; NCT02224573). All participants who did not immediately enter the OLE study tapered investigational medicinal product (IMP) (10% per day over 10 days). However, the taper period could be interrupted if the participant wished to enter the OLE study within a 7-day timeframe. Participants who down-titrated IMP returned for an end of taper period visit (Day 109). Participants who did not enter the OLE study or who withdrew prematurely had a safety follow-up visit 28 days later (Day 137).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant and/or parent(s)/legal representatives were willing and able to give informed assent/consent for participation in the study.
* Participant and his or her caregivers were willing and able (in the investigator's opinion) to comply with all study requirements.
* Participant was male or female aged between 2 and 55 years (inclusive).
* Participant had a documented history of LGS. This included written documentation of having met electroencephalogram (EEG) diagnostic criteria during the participant's history and evidence of at least 1 type of generalized seizure, including drop seizures (atonic, tonic, tonic-clonic or myoclonic) for at least 6 months.
* Participant had a history of slow (<3.0 hertz [Hz]) spike-and-wave pattern in an EEG prior to the enrollment into the baseline period.
* Participant had at least 2 drop seizures each week during the first 28 days of the baseline period.
* Participant was refractory; that is having documented failures on more than 1 antiepileptic drug (AED).
* Participant was taking 1 or more AEDs at a dose which had been stable for at least 4 weeks prior to screening.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation [VNS]) were stable for 4 weeks prior to screening and the participant was willing to maintain a stable regimen throughout the study. The ketogenic diet and VNS treatments were not counted as an AED.
* Participant and/or parent(s)/legal representatives were willing to allow his or her primary care practitioner and consultant to be notified of participation in the study.
* Participant completed his or her interactive voice response (IVRS) telephone diary on at least 25 days of the baseline period.

Key Exclusion Criteria:

* Etiology of participant's seizures was a progressive neurologic disease. Participants with tuberous sclerosis were not excluded from study participation, unless there was a progressive tumor.
* Participant had an anoxic episode requiring resuscitation within 6 months of screening.
* Participant had clinically significant unstable medical conditions other than epilepsy.
* Participant had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to screening or randomization, other than epilepsy.
* Participant had a history or presence of alcohol or substance abuse within the last 2 years prior to the study or daily consumption of 5 or more alcohol-containing beverages.
* Participant was currently using or had in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to study entry and was unwilling to abstain for the duration of the study.
* Participant had a history of symptoms (for example, dizziness, light-headedness, blurred vision, palpitations, weakness, syncope) related to a drop in blood pressure due to postural changes.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP, such as sesame oil.
* Female participant was of child bearing potential or male participant's partner was of child bearing potential; unless willing to ensure that they or their partner used a highly effective method of contraception for the duration of the study and for 3 months thereafter.
* Female participant was pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the study and for 3 months thereafter.
* Participant had been part of a clinical study involving another IMP in the previous 6 months.
* Patient had significantly impaired hepatic function at screening (Day -28) or randomization (Day 1), defined as any of the following: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); ALT or AST > 3 × ULN and total bilirubin > 2 × ULN or international normalized ratio (INR) > 1.5; ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%). This criterion could only be confirmed once the laboratory results were available; participants randomized into the study who were later found not to meet this criterion were withdrawn from the study.
* Any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale in the last month or at screening.
* Participant was unwilling to abstain from donation of blood during the study.
* Participant planned to travel outside his or her country of residence during the study.
* Participant had previously randomized into the study.
* Participant was taking more than 4 concurrent AEDs.
* Participant had taken corticotropins in the 6 months prior to screening.
* Participant was currently taking long-term systemic steroids (excluding inhaled medication for asthma treatment) or any other daily medication known to exacerbate epilepsy. An exception was made of prophylactic medication, for example, idiopathic nephrotic syndrome or asthma.
* Participant was taking felbamate, and he or she had been taking it for less than 1 year prior to screening.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (19):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Hartford, Connecticut
  - Orlando, Florida
  - Augusta, Georgia
  - Boise, Idaho
  - Rochester, Minnesota
  - Buffalo, New York
  - New York, New York
  - Clemmons, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - York, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Fort Worth, Texas
  - Charlottesville, Virginia
- Paris, France
- Spain (5):
  - Barcelona
  - Madrid
  - Pamplona
  - Seville
  - Valencia
- United Kingdom (3):
  - Edinburgh
  - Glasgow
  - London

REFERENCES:
- [Result] Devinsky O, Patel AD, Cross JH, Villanueva V, Wirrell EC, Privitera M, Greenwood SM, Roberts C, Checketts D, VanLandingham KE, Zuberi SM; GWPCARE3 Study Group. Effect of Cannabidiol on Drop Seizures in the Lennox-Gastaut Syndrome. N Engl J Med. 2018 May 17;378(20):1888-1897. doi: 10.1056/NEJMoa1714631. PMID 29768152
- [Derived] Specchio N, Auvin S, Greco T, Lagae L, Nortvedt C, Zuberi SM. Clinically Meaningful Reduction in Drop Seizures in Patients with Lennox-Gastaut Syndrome Treated with Cannabidiol: Post Hoc Analysis of Phase 3 Clinical Trials. CNS Drugs. 2025 Oct;39(10):1025-1036. doi: 10.1007/s40263-025-01201-8. Epub 2025 Aug 7. PMID 40775196
- [Derived] Auvin S, Nortvedt C, Fuller DS, Sahebkar F. Seizure-free days as a novel outcome in patients with Lennox-Gastaut syndrome: Post hoc analysis of patients receiving cannabidiol in two randomized controlled trials. Epilepsia. 2023 Jul;64(7):1812-1820. doi: 10.1111/epi.17618. Epub 2023 Apr 28. PMID 37052803
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- [Derived] Privitera M, Bhathal H, Wong M, Cross JH, Wirrell E, Marsh ED, Mazurkiewicz-Beldzinska M, Villanueva V, Checketts D, Knappertz V, VanLandingham K. Time to onset of cannabidiol (CBD) treatment effect in Lennox-Gastaut syndrome: Analysis from two randomized controlled trials. Epilepsia. 2021 May;62(5):1130-1140. doi: 10.1111/epi.16878. Epub 2021 Apr 2. PMID 33797076
- [Derived] Perry MS. Don't Fear the Reefer-Evidence Mounts for Plant-Based Cannabidiol as Treatment for Epilepsy. Epilepsy Curr. 2019 Mar-Apr;19(2):93-95. doi: 10.1177/1535759719835671. PMID 30955420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The dose levels of 10 and 20 milligram (mg) per kilogram (kg) per day (mg/kg/day) were recommended by the Data Safety Monitoring Committee (DSMC) of study GWEP1332 Part A (NCT02091206) after assessment of safety and pharmacokinetic data. Participants of GWEP1414 were not enrolled until the DSMC had reviewed the safety data of GWEP1332 Part A.
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received GWP42003-P 20 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the open-label extension (OLE) study, the maintenance period was followed by a 10-day taper (10% per day) period.
- Placebo: Participants received placebo (0 mg/milliliter [mL] cannabidiol [CBD]), volume matched to 1 of the 2 dose levels (10 or 20 mg/kg/day), administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 7 to 11 days according to the matched investigational medicinal product (IMP) group (7 or 11 days for the 10 or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period.
Period: Overall Study
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | Placebo
Started | 76 | 73 | 76
Safety Analysis Set (Received at least 1 dose of IMP; analyzed as per actual treatment received.) | 82 (Six participants assigned to the 10 mg/kg/day dose were included in the 20 mg/kg/day group.) | 67 (Six participants assigned to the 10 mg/kg/day dose were included in the 20 mg/kg/day group.) | 76
Intent to Treat (ITT) Analysis Set (Received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement.) | 76 | 73 | 76
Completed | 67 | 71 | 74
Not Completed | 9 | 2 | 2
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Met Withdrawal Criteria | 1 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Withdrawn by Investigator | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set: Received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement. Participants were analyzed according to the treatment group to which they were randomized.
Groups:
- GWP42003-P 20 mg/kg/Day Dose-ITT Analysis Set: Participants received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement; analyzed according to the treatment group to which they were randomized (GWP42003-P 20 mg/kg/day).
- GWP42003-P 10 mg/kg/Day Dose-ITT Analysis Set: Participants received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement; analyzed according to the treatment group to which they were randomized (GWP42003-P 10 mg/kg/day).
- Placebo-ITT Analysis Set: Participants received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement; analyzed according to the treatment group to which they were randomized (Placebo).
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 20 mg/kg/Day Dose-ITT Analysis Set | GWP42003-P 10 mg/kg/Day Dose-ITT Analysis Set | Placebo-ITT Analysis Set | Total
Number analyzed (Participants) | 76 | 73 | 76 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (10.8) | 15.4 (9.5) | 15.3 (9.3) | 15.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 32 | 96
  Male | 45 | 40 | 44 | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline In Drop Seizure Frequency During The Treatment Period
Description: Drop seizures were recorded by the participant or caregiver using an interactive voice response system (IVRS) diary. Drop seizures were defined as the subset of tonic-clonic, tonic or atonic seizures that were reported as drop seizures in the IVRS. Percentage change from baseline was calculated as: ([frequency during the treatment period - frequency during baseline]/frequency during baseline) x 100. The frequency during each period was based on 28-day averages and calculated as: (number of seizures in the period/number of reported days in the IVRS period) x 28. Baseline included all available data prior to Day 1 (28-day average). Negative percentages show an improvement from baseline.
Time Frame: Baseline to End of Treatment (EOT) (Day 99) or Early Termination (ET)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: percentage change
Groups:
- Placebo: Participants received placebo (0 mg/mL CBD), volume matched to 1 of the 2 dose levels (10 or 20 mg/kg/day), administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 7 to 11 days according to the matched IMP group (7 or 11 days for the 10 or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period.
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 76 | 73 | 76
percentage change | -41.86 [-72.4 to -1.3] | -37.16 [-63.8 to -5.6] | -17.17 [-37.1 to 0.9]
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0047, Wilcoxon rank-sum test; Median Difference (Final Values) = -21.57, 95% CI 2-sided [-34.79 to -6.67] — Calculated using the Hodges-Lehmann approach
Statistical Analysis 2: Comparison: GWP42003-P 10 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0016, Wilcoxon rank-sum test; Median Difference (Final Values) = -19.19, 95% CI 2-sided [-31.24 to -7.69] — Calculated using the Hodges-Lehmann approach

2. Secondary Outcome: Number Of Participants With A ≥50% Reduction From Baseline In Drop Seizure Frequency During The Treatment Period
Description: Drop seizures were recorded by the participant or caregiver using an IVRS diary. Drop seizures included the subset of tonic-clonic, tonic, or atonic seizures that were reported as drop seizures in IVRS. Percentage change from baseline was calculated as per the primary outcome measure.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 76 | 73 | 76
Participants | 30 | 26 | 11
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — Calculated using a Cochran-Mantel-Haenszel (CMH) test stratified by age group (2-5, 6-11, 12-17 and 18-55 years); Odds Ratio (OR) = 3.85, 95% CI 2-sided [1.75 to 8.47]
Statistical Analysis 2: Comparison: GWP42003-P 10 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel — Calculated using a CMH test stratified by age group (2-5, 6-11, 12-17 and 18-55 years); Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.47 to 7.26]

3. Secondary Outcome: Percentage Change From Baseline In Total Seizure Frequency During The Treatment Period
Description: Total seizures included the sum of all seizures (tonic-clonic, tonic, atonic, clonic, myoclonic, countable partial, other partial, and absence seizures) recorded by the participant or caregiver using an IVRS diary. Percentage change from baseline was calculated as per the primary outcome measure. Negative percentages show an improvement from baseline.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 76 | 73 | 76
percentage change | -38.40 [-64.6 to -0.7] | -36.44 [-64.5 to -10.8] | -18.47 [-39.0 to 0.5]
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0091, Wilcoxon rank-sum test; Median Difference (Final Values) = -18.76, 95% CI 2-sided [-31.80 to -4.43] — Calculated using the Hodges-Lehmann approach
Statistical Analysis 2: Comparison: GWP42003-P 10 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0015, Wilcoxon rank-sum test; Median Difference (Final Values) = -19.47, 95% CI 2-sided [-30.37 to -7.47] — Calculated using the Hodges-Lehmann approach

4. Secondary Outcome: Subject/Caregiver Global Impression Of Change (S/CGIC) Assessment
Description: The S/CGIC was used to assess the participant's overall condition on a 7-point scale, using the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse" (1 = very much improved; 7 = very much worse). On Day 1 (prior to starting IMP), the caregiver was asked to write a brief description of the participant's overall condition as a memory aid for the S/CGIC questionnaire at subsequent visits. If both a CGIC and SGIC were completed then the CGIC was used; if only a CGIC was completed then the CGIC was used; if only a SGIC was completed then the SGIC was used. Last visit for endpoints assessed at clinic visits was defined as the last scheduled visit (not including the end of taper or safety follow-up visits) at which participant's last evaluation was performed.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 75 | 73 | 75
Participants
  Very Much Improved | 6 | 9 | 1
  Much Improved | 15 | 14 | 8
  Slightly Improved | 22 | 25 | 24
  No Change | 25 | 21 | 35
  Slightly Worse | 6 | 3 | 4
  Much Worse | 1 | 1 | 3
  Very Much Worse | 0 | 0 | 0
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0439, Regression, Logistic; Ordinal logistic regression model with treatment group as a fixed factor; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.02 to 3.30] — Odds of participant recording a lower score (improvement) on a continuous scale
Statistical Analysis 2: Comparison: GWP42003-P 10 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0020, Regression, Logistic; Ordinal logistic regression model with treatment group as a fixed factor; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.41 to 4.66] — Odds of participant recording a lower score (improvement) on a continuous scale

ADVERSE EVENTS:
Time Frame: Day 1 through Day 137 (Safety Follow-up)
Description: Safety Analysis Set: Received at least 1 dose of IMP; analyzed as per actual treatment received. Six participants who were assigned to the GWP42003-P 10 mg/kg/day dose received dosing schedules for GWP42003-P 20 mg/kg/day. For safety analyses, these participants were assigned to the GWP42003-P 20 mg/kg/day group.
Groups:
- GWP42003-P 20 mg/kg/Day Dose-Safety Analysis Set; GWP42003-P 10 mg/kg/Day Dose-Safety Analysis Set: Participants received at least 1 dose of IMP; analyzed as per actual treatment received. Six participants who were assigned to the GWP42003-P 10 mg/kg/day dose received dosing schedules for GWP42003-P 20 mg/kg/day. For safety analyses, these participants were assigned to the GWP42003-P 20 mg/kg/day group.
- Placebo-Safety Analysis Set: Participants received at least 1 dose of IMP; analyzed as per actual treatment received.
Arm/Group | GWP42003-P 20 mg/kg/Day Dose-Safety Analysis Set | GWP42003-P 10 mg/kg/Day Dose-Safety Analysis Set | Placebo-Safety Analysis Set
Serious Adverse Events (participants affected / at risk) | 13/82 | 13/67 | 8/76
Other Adverse Events (participants affected / at risk) | 63/82 | 36/67 | 40/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose-Safety Analysis Set (N=82) | GWP42003-P 10 mg/kg/Day Dose-Safety Analysis Set (N=67) | Placebo-Safety Analysis Set (N=76)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Device malfunction (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Investigation (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 4 | 7 | 3
Convulsion (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose-Safety Analysis Set (N=82) | GWP42003-P 10 mg/kg/Day Dose-Safety Analysis Set (N=67) | Placebo-Safety Analysis Set (N=76)
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 6
Vomiting (Gastrointestinal disorders) | 10 | 4 | 9
Pyrexia (General disorders) | 9 | 6 | 12
Fatigue (General disorders) | 8 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 11 | 11
Nasopharyngitis (Infections and infestations) | 9 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 21 | 11 | 6
Somnolence (Nervous system disorders) | 25 | 14 | 4
Lethargy (Nervous system disorders) | 5 | 3 | 2
Convulsion (Nervous system disorders) | 5 | 2 | 7
Headache (Nervous system disorders) | 5 | 2 | 3
Irritability (Psychiatric disorders) | 4 | 6 | 2
Insomnia (Psychiatric disorders) | 4 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days